CLINICAL TRIAL: NCT06750718
Title: Virtual Reality Neck-based Sensorimotor Training Versus Comprehensive Sensorimotor Training in Mechanical Neck Pain
Brief Title: Innovative Rehabilitation: Integrating VR-Based Sensorimotor Training Into Comprehensive Neck Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal Abd-Elmaboud Maghraby, Assistant lecturer at the Faculty of Physical Therapy, Department of Physical Therapy for Musculoskeletal Disorders and Surgeryز, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005274
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Non Specific Neck Pain
Keywords: Virtual Reality (VR); Non specific Neck Pain (NSNP); Neck-based Training Sensorimotor Training; Sensorimotor Training

STUDY DESIGN:
Intervention Model Description: Fifty patients with mechanical neck pain patients will be randomly allocated into 2 equal groups; group (A) received VR neck-based sensorimotor training only, group (B) received comprehensive sensorimotor training only. (Parallel Group Two-Armed Comparative Randomized Controlled Trial)
Who Masked: Outcomes Assessor
Masking Description: A blinded researcher will assess the patients during the trial, blinding will not be feasible for participants or therapists due to the layout of the VR therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The virtual reality group will engage in targeted cervical sensorimotor training through VR Oculus Quest 2 (OQ2)
  Interventions: Device: Virtual Reality (VR)
- Comprehensive Sensorimotor Training (Active Comparator): An exercise program consisting of Cervical JPSM, Cervical movement sense, and Oculomotor control exercises.
  Interventions: Other: Comprehensive Sensorimotor Training

INTERVENTIONS:
Device: Virtual Reality (VR) — Oculus Quest 2 (OQ2) advanced 256 GB all-in-one virtual reality headset, Wi-Fi will be used.
  Other Names: Oculus Quest 2 (OQ2)
  Arms: Virtual Reality
Other: Comprehensive Sensorimotor Training — An exercise program consisting of Cervical JPSM, Cervical movement sense, and Oculomotor control exercises.
  Arms: Comprehensive Sensorimotor Training

SUMMARY:
The research aims to treat chronic non-specific neck pain using virtual reality (VR) technologies with sensory-motor training. Chronic neck pain is widespread and highly prevalent in Egyptian society due to many factors, such as sitting for long periods in front of a computer or smartphone, which leads to a decline in productivity at work and a constant feeling of fatigue. This problem is considered one of the widespread health problems that affect individuals of all ages and greatly affect their daily lives.

This project was chosen based on the growing awareness of the need to search for innovative solutions to this health problem that hinders productivity and affects the general comfort of individuals.

The reserch aims to integrate sensory-motor therapy with virtual reality, which helps patients improve movement and flexibility and reduce pain. It does this by simulating exciting interactive environments that engage their attention and help them relieve pain away from traditional treatment methods.

DETAILED DESCRIPTION:
Virtual reality, a novel form of technology, is gaining attention in the medical field for its potential to aid inpatient rehabilitation. This experience will immerse the patient in an interactive and engaging journey. Virtual reality feedback can assist patients with chronic musculoskeletal pain by offering them various sensory and motor tasks to enhance their postural control.

Moreover, virtual reality offers a distracting experience that aids in reducing patients' pain and emotional distress. Using a specialized device on their head (Head-mounted device) (HMD) or screen, patients can participate in computer-based exercises as part of virtual reality physical therapy.

Combining virtual reality with comprehensive sensorimotor training can be beneficial in treating chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty patients diagnosed with mechanical neck pain between 18- and 40 years old with mechanical neck pain.
2. Patients with pain intensity scores (>3) on the visual analog scale (VAS; 0-100mm) for an average of three weeks before the study.
3. Neck Disability Index (NDI) scoring 20%-60% (>6) (moderate to severe disability).

Exclusion Criteria:

1. Any history of lower extremity or spine trauma or surgery, recognized and observable spinal deformity, neurological disorders, cervical fracture/dislocation, whiplash injuries, neurological/cardiovascular/respiratory disorders affecting patients' physical performance, or inability to provide informed consent.
2. Benign paroxysmal positional vertigo (BPPV), as confirmed by the Dix Hallpike test.
3. Pregnancy.
4. Patients who had received physical therapy interventions for neck pain within three months preceding the study were also ineligible for participation and were excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of pain intensity (VAS) | Before Treatment and after 6 weeks of treatment
  Asking the patient to put a horizontal mark on a continuous 10 cm line that represents his/her pain intensity, ranging from zero, which indicates no pain, or 29 discomfort to 10, which indicates the worst possible pain he could feel.
Measurement of disability due to neck pain (NDI) | Before Treatment and after 6 weeks of treatment
  The patient will complete a condition-specific functional status questionnaire with 10 items. The NDI consists of 10 domains-pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleep, and recreation-designed to assess the level of disability in patients with neck pain. Patients self-report their level of function/disability in each domain, after which a composite score is calculated.
Cervical proprioception and neck reposition sense | Before Treatment and after 6 weeks of treatment
  Cervical joint position error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability.
Eye Movement Control (Gaze Stability) | Before Treatment and after 6 weeks of treatment
  The Dynamic Visual Acuity (DVA) test is used for assessing gaze stability.
Cervical range of motion (ROM) | Before Treatment and after 6 weeks of treatment
  Cervical ROM results were calculated by averaging the three best values from each direction
Cervical kinematics: Peak velocity (V peak /sec) | Before Treatment and after 6 weeks of treatment
  Calculated as the maximal angular velocity, from motion initiation to target hit.
Cervical kinematics: Mean velocity (V mean /sec) | Before Treatment and after 6 weeks of treatment
  The mean angular velocity angular velocity, from motion initiation to target hit
Cervical kinematics: Time to peak velocity percentage (TTP%) | Before Treatment and after 6 weeks of treatment
  The time from motion initiation to peak velocity moment, as a percentage of total movement time, representing the ratio between the acceleration to deceleration phase in the velocity profile
Cervical kinematics: Static head stability (sway) | Before Treatment and after 6 weeks of treatment
  The sway in pitch and yaw from the mid-position and calculated in terms of 3D mean and standard deviation amplitude
Cervical kinematics: Head movement accuracy | Before Treatment and after 6 weeks of treatment
  Motion accuracy was defined as the difference between the target position and the participant's head location. This difference (target position- player's head position)

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer Maghraby, MSc, Principal Investigator — Assistant Lecturer
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Physical Therapy, Cairo